CLINICAL TRIAL: NCT02602366
Title: The Quatro Study: Acceptability Study of (Placebo) Vaginal Delivery Forms for Preventing HIV and Unintended Pregnancy Among Young Women in Zimbabwe and South Africa
Brief Title: The Quatro Study: Acceptability Study of (Placebo) Vaginal Delivery Forms for Preventing HIV and Unintended Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CONRAD (Other)
Collaborators: RTI International (Other); UZ-UCSF Collaborative Research Programme (Other); Match Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Quatro
Record Dates: First submitted 2015-11-09; First posted 2015-11-11 (Estimated); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: HIV; Contraception
Keywords: HIV; DCE; MPT; Microbicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Month 1 (Other): In a cross-over design, women will be randomized to a sequence of product use. Each product will be tested by every participant for 1 month in a 4-period cross-over design.
  Interventions: Other: HEC Placebo Gel; Other: Placebo Vaginal Insert; Other: Placebo Vaginal Film; Other: Placebo Intravaginal ring (IVR)
- Month 2 (Other): In a cross-over design, women will be randomized to a sequence of product use. Each product will be tested by every participant for 1 month in a 4-period cross-over design.
  Interventions: Other: HEC Placebo Gel; Other: Placebo Vaginal Insert; Other: Placebo Vaginal Film; Other: Placebo Intravaginal ring (IVR)
- Month 3 (Other): In a cross-over design, women will be randomized to a sequence of product use. Each product will be tested by every participant for 1 month in a 4-period cross-over design.
  Interventions: Other: HEC Placebo Gel; Other: Placebo Vaginal Insert; Other: Placebo Vaginal Film; Other: Placebo Intravaginal ring (IVR)
- Month 4 (Other): In a cross-over design, women will be randomized to a sequence of product use. Each product will be tested by every participant for 1 month in a 4-period cross-over design.
  Interventions: Other: HEC Placebo Gel; Other: Placebo Vaginal Insert; Other: Placebo Vaginal Film; Other: Placebo Intravaginal ring (IVR)

INTERVENTIONS:
Other: HEC Placebo Gel
Other: Placebo Vaginal Insert
Other: Placebo Vaginal Film
Other: Placebo Intravaginal ring (IVR)

SUMMARY:
The purpose of The Quatro Study is to assess the acceptability, preferences, user experience and effect on sexual behavior of four different vaginal microbicide or multi-purpose technology (MPT) delivery forms, using placebo products in 18-30 year old African women: rapidly disintegrating vaginal insert, intravaginal ring (IVR), film and gel. The study also examines adherence to the dosage forms through objective markers, developed for each dosage form prior to the commencement of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-30
* In good health, as determined by the site Investigator or designee based on clinical history
* Willing and able to comply with study procedures and attend monthly follow-up visits
* Willing and able to provide informed consent
* Fluent in one of the languages being used in the study (English, Shona or Zulu)
* Not intending to travel or move out of the research catchment area for the next 6 months
* Sexually active defined by vaginal intercourse with a male at least 4 times per month in the past 3 months and plan to be sexually active during the study duration

Exclusion Criteria:

* HIV positive
* Pregnant, or intention to become pregnant during the clinical study
* Prior participation in any HIV-prevention or MPT product demonstration study or clinical trial
* Any current or historical health (including vaginal or genitourinary conditions) or psychological issues that the site Investigator or his/her designee determines should exclude the potential participant

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 422 (Actual)
Dates: Start 2016-06-06 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in ratings and relative preference rankings of four vaginal delivery forms | Baseline, Month 1, Month 2, Month 3, Month 4, Month 5

SECONDARY OUTCOMES:
Attributes least and most favored for the vaginal delivery forms as measured by discreet choice experiment | Month 5
Adherence assessed by self report via questionnaire | Baseline, Month 1, Month 2, Month 3, Month 4, Month 5
Adherence assessed by objective biomarkers, utilizing antibodies, tagged recombinant proteins, biochemical assays and/or spectroscopy | Baseline, Month 1, Month 2, Month 3, Month 4, Month 5

CONTACTS AND LOCATIONS:
Overall Officials: Jill Schwartz, MD, MPH, Principal Investigator — CONRAD
Locations (2):
- MatCH Research, Durban, South Africa
- The University of Zimbabwe-University of California San Francisco Collaborative Research Program (UZ-UCSF), Harare, Zimbabwe